CLINICAL TRIAL: NCT02121158
Title: CSP #592 - Efficacy and Safety of ICD Implantation in the Elderly
Brief Title: Efficacy and Safety of Implantable Cardioverter-Defibrillator (ICD) Implantation in the Elderly
Acronym: I-70
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results of the pilot were not enough to justify the extension of the pilot. Results presented are from pilot.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 592
Record Dates: First submitted 2014-04-16; First posted 2014-04-23 (Estimated); Results first posted 2022-01-20 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cardiomyopathy; Coronary Artery Disease; Congestive Heart Failure; Myocardial Infarction
Keywords: CSP 592; ICD; cardiovascular; heart; aging; chronic diseases; multi-site trial; investigational device; cardiomyopathy; coronary artery disease; congestive heart failure; myocardial infarction; I-70; I70; elderly; defibrillator
MeSH Terms: conditions — Cardiomyopathies; Coronary Artery Disease; Heart Failure; Myocardial Infarction; Chronic Disease | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 1 (Other): ICD implantation in addition to Optimal Medical Therapy
  Interventions: Device: Implantable Cardioverter Defibrillator
- 2 (Active Comparator): Optimal Medical Therapy
  Interventions: Other: Optimal Medical Therapy

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator — The ICD and lead(s) will be FDA-approved.
  Arms: 1
Other: Optimal Medical Therapy — Guidance on lifestyle modification, exercise training, and disease management including review of American Heart Association (AHA) Guidelines for Primary Prevention of Cardiovascular Disease and Stroke.
  Arms: 2

SUMMARY:
The overall aim of this trial is to study the safety and efficacy of ICD implantation as a primary prevention strategy of sudden cardiac death in patients 70 years and older. This study will assess the many competing factors involved with ICD implantation including 1) the impact on mortality, especially in the context of a declining rate of sudden death with advanced age, 2) the tolerability of the powerful therapeutic action of the device, and 3) the impact on quality of life.

DETAILED DESCRIPTION:
The overall aim of this trial is to study the safety and efficacy of ICD implantation as a primary prevention strategy of sudden cardiac death (SCD) in patients 70 years and older. In particular, this study is designed to determine the comparative effectiveness of ICD, in addition to optimal medical therapy (OMT), in reducing all-cause mortality, versus OMT alone; OMT includes standard intervention for chronic heart failure patients, i.e. lifestyle modification, disease management, adoption of healthy diet and exercise practices, etcetera. One particularly important secondary objective is to assess treatment efficacy under the conditions of high versus low co-morbidity burden.

Participants will be randomized (1:1 ratio) to ICD + OMT or OMT alone, and stratified by participating site and co-morbidity level (Charlson score <3 versus 3+). Acute treatment visits will occur as clinically indicated and per local convention; follow-up will occur 1-4 months post-randomization (all participants), and not sooner than 30 days - and not later than 120 days post-implantation (ICD arm); regular follow-up will occur at 6 month intervals post-randomization until study close (all participants). All follow-up will be conducted centrally. Neither the participant nor treating clinician will be masked to treatment.

Primary Objective:

The primary objective of this study is to determine if a primary prevention strategy with ICD implantation in addition to optimal medical therapy (OMT) is effective in reducing all-cause mortality compared to OMT alone in patients 70 years of age and older who are eligible for ICD therapy according to current Centers for Medicare & Medicaid Services (CMS) criteria.

Primary Hypothesis:

The primary hypothesis of this study is that implantation of an ICD plus optimal medical therapy will reduce all-cause mortality in patients 70 years of age and older versus optimal medical therapy alone.

Secondary Objectives:

1. One secondary objective of this study is to ascertain whether age, co-morbidity burden, or age and burden together, are determinants in mortality outcomes in the OMT versus ICD + OMT group.
2. An additional secondary objective of the study is to determine the effect of ICD implantation plus optimal medical therapy on quality of life among elderly patients compared with optimal medical therapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. 70 years of age or older
2. Eligible for ICD implementation according to the CMS criteria for primary prevention by one of the following conditions:

   1. Documented prior MI and a measured left ventricular ejection fraction (LVEF) <=30% (includes New York Heart Association [NYHA] class I, II, or III)
   2. Coronary artery disease with a documented prior MI, a measured left ventricular ejection fraction <=35%, and inducible, sustained ventricular tachycardia (VT) or ventricular fibrillation (VF) at electrophysiology (EP) study
   3. Ischemic dilated cardiomyopathy (IDCM), documented prior MI, NYHA class II and III heart failure, and measured LVEF <=35%
   4. Non-ischemic dilated cardiomyopathy (NIDCM) > 3 months, NYHA Class II and III heart failure, and measured LVEF <=35%
3. Stable condition on Optimal Medical Therapy
4. Able and willing to provide informed consent to participate in this study

Exclusion Criteria:

1. Enrolled in or planning to enroll in a conflicting trial
2. Receiving a bi-ventricular ICD device
3. New York Heart Association class IV heart failure
4. Cardiogenic shock or symptomatic hypotension while in stable baseline rhythm,
5. Coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) within the past 3 months
6. An MI within the past 40 days
7. Clinical symptoms or findings that would make them a candidate for coronary revascularization
8. Irreversible brain damage from pre-existing cerebral disease
9. Any disease other than cardiac disease (e.g. cancer, uremia, liver failure), associated with a likelihood of survival less than 1 year
10. Circumstance that would prevent completion of the trial and follow-up activities, including medical condition

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Singh, MD, Study Chair — Washington DC VA Medical Center, Washington, DC
Locations (5):
- United States (5):
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singh SN, Wininger M, Raitt M, Adabag S, Moore H, Rottman JN, Scrymgeour A, Zhang J, Zheng K, Guarino P, Kyriakides TC; I-70 Study Group; Johnson G, Williams A, Beed A, MacMurdy K, Saavedra P. Efficacy and safety of implantable cardioverter-defibrillator implantation in the elderly-The I-70 Study: A randomized clinical trial. Heart Rhythm O2. 2024 Apr 27;5(6):365-373. doi: 10.1016/j.hroo.2024.04.010. eCollection 2024 Jun. PMID 38984364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at six Department of Veterans Affairs Medical Centers (VAMCs). Recruitment start: 8/6/2015 (4) 9/25/2015 (1) and 10/29/2015 (1). Recruitment terminated: 12/6/2016 (1) and 12/5/2019 (5).
Pre-assignment Details: None: Study design did not include significant events that occur after participant enrollment: no run-in phase, nor wash-out.
Groups:
- Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD): Guidance on lifestyle modification, exercise training, and disease management including review of American Heart Association (AHA) Guidelines for Primary Prevention of Cardiovascular Disease and Stroke + FDA-Approved implantable cardioverter defibrillator and leads.
Period: Overall Study
Arm/Group | Optimal Medical Therapy | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD)
Started | 85 | 82
Completed | 85 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimal Medical Therapy | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD) | Total
Number analyzed (Participants) | 85 | 82 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 85 | 82 | 167
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 84 | 81 | 165
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 73 | 67 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85 | 82 | 167
New York Heart Association Class: I [Count of Participants; unit: Participants] — Participants were evaluated for their NYHA class level according to the criteria adapted in Dolgin M, 1994 (Dolgin M Association NYH, Fox AC, Gorlin R, Levin RI, New York Heart Association. Criteria Committee. Nomenclature and criteria for diagnosis of diseases of the heart and great vessels. 9th ed. Boston, MA: Lippincott Williams and Wilkins; March 1, 1994.).
  Class I = No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Participants | 2 | 4 | 6
New York Heart Association Class: II [Count of Participants; unit: Participants] — Participants were evaluated for their NYHA class level according to the criteria adapted in Dolgin M, 1994 (Dolgin M Association NYH, Fox AC, Gorlin R, Levin RI, New York Heart Association. Criteria Committee. Nomenclature and criteria for diagnosis of diseases of the heart and great vessels. 9th ed. Boston, MA: Lippincott Williams and Wilkins; March 1, 1994.).
  Class II = Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Participants | 62 | 58 | 120
New York Heart Association Class: III [Count of Participants; unit: Participants] — Participants were evaluated for their NYHA class level according to the criteria adapted in Dolgin M, 1994 (Dolgin M Association NYH, Fox AC, Gorlin R, Levin RI, New York Heart Association. Criteria Committee. Nomenclature and criteria for diagnosis of diseases of the heart and great vessels. 9th ed. Boston, MA: Lippincott Williams and Wilkins; March 1, 1994.).
  Class III = Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Participants | 21 | 20 | 41
New York Heart Association Class: IV [Count of Participants; unit: Participants] — Participants were evaluated for their NYHA class level according to the criteria adapted in Dolgin M, 1994 (Dolgin M Association NYH, Fox AC, Gorlin R, Levin RI, New York Heart Association. Criteria Committee. Nomenclature and criteria for diagnosis of diseases of the heart and great vessels. 9th ed. Boston, MA: Lippincott Williams and Wilkins; March 1, 1994.).
  Class IV = Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: All-cause mortality
Time Frame: Through study completion, starting from consent/baseline: average of 31 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Optimal Medical Therapy | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD)
Number analyzed (Participants) | 85 | 82
Participants | 23 | 20

2. Secondary Outcome: Quality of Life - Minnesota Living With Heart Failure Questionnaire
Description: Minnesota Living with Heart Failure questionnaire. MLHF scoring: 0 points = Best QOL, 105 points = Worst QOL.
Time Frame: Measured at 12-months post-randomization
Population: Analysis population differs from total number of study participants due to non-completion of the 12-month study visit, explained by either patient expiry or missed visit.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Optimal Medical Therapy | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD)
Number analyzed (Participants) | 62 | 63
score on a scale | 11 [6.0 to 26.5] | 13 [5.0 to 37.0]

3. Secondary Outcome: Sudden Cardiac Death
Description: Sudden Cardiac Death
Time Frame: Through study completion, starting from consent/baseline: average of 31 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Optimal Medical Therapy | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD)
Number analyzed (Participants) | 85 | 82
Participants | 5 | 3

4. Secondary Outcome: All-cause Hospitalization
Description: Number of participants hospitalized during study follow-up
Time Frame: Through study completion, starting from consent/baseline: average of 31 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Optimal Medical Therapy | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD)
Number analyzed (Participants) | 85 | 82
Participants | 61 | 60
Statistical Analysis 1: Comparison: Optimal Medical Therapy vs Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD); Test type: Equivalence — Unadjusted; p = 0.7457, Cox Proportional Hazards; Hazard Ratio (HR) = 0.915, 95% CI 2-sided [0.534 to 1.568]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were monitored from consent/baseline through 30 days after study exit, an average of 31 months. Non-Serious Adverse Events were monitored from consent/baseline through 30 days (30 days only, i.e. 30 days past consent [OMT arm] or 30 days past implantation [ICD arm]), i.e. 30 days for all participants.
Arm/Group | Optimal Medical Therapy | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD)
All-Cause Mortality (participants affected / at risk) | 23/85 | 20/82
Serious Adverse Events (participants affected / at risk) | 67/85 | 62/82
Other Adverse Events (participants affected / at risk) | 1/85 | 6/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optimal Medical Therapy (N=85) | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD) (N=82)
Bleeding (Metabolism and nutrition disorders) | 0 | 1
Infection (ICD) (Infections and infestations) | 1 | 0
Infection (other) (Infections and infestations) | 26 | 32
Lead Alteration (Product Issues) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 12 | 8
Atrial fibrillation / Atrial flutter (Cardiac disorders) | 9 | 2
Stroke (Nervous system disorders) | 2 | 3
HF Complication (Cardiac disorders) | 57 | 54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optimal Medical Therapy (N=85) | Optimal Medical Therapy + Implantable Cardioverter Defibrillator (OMT + ICD) (N=82)
Painful implant site (General disorders) | 0 | 6
New dizziness (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT02121158/Prot_SAP_ICF_000.pdf